CLINICAL TRIAL: NCT06225570
Title: Randomized Controlled Trial of Weekly Oral Isotretinoin vs. Oral Tetracyclines for the Treatment of Moderate Acne Vulgaris
Brief Title: Weekly Isotretinoin vs Tetracycline for Moderate Acne
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00131877
Record Dates: First submitted 2023-12-14; First posted 2024-01-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Acne Vulgaris
Keywords: moderate acne vulgaris; isotretinoin
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin; Tetracycline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Isotretinoin (Experimental): Weekly isotretinoin (at 1-1.5 mg/kg per week) dose preceded by a 5-day daily loading dose (0.5-1 mg/kg/day). The weekly dose will be given once a week for 4 months.
  Interventions: Drug: Isotretinoin
- Tetracycline (Active Comparator): Daily oral doxycycline (weight-based dosing with maximum dose 200mg daily) or other tetracycline class antibiotic for a 4-month treatment period.
  Interventions: Drug: Tetracycline

INTERVENTIONS:
Drug: Isotretinoin — This arm aims to study the effectiveness, side effects and patient satisfaction of taking isotretinoin on a weekly basis as opposed to current standard daily dosing.
  Arms: Isotretinoin
Drug: Tetracycline — This arm aims to serve as the comparison group. Tetracycline antibiotics are the current standard of care for the treatment of moderate acne.
  Arms: Tetracycline

SUMMARY:
In the effort to find better treatments for Moderate Acne, which often relies on long-term antibiotic use, researchers are exploring alternative options. While Isotretinoin, a Vitamin A derivative, is highly effective for severe acne, its side effects limit its use for milder cases. A recent study from our institution investigated a new approach: weekly Isotretinoin dosing. The results were promising, with acne improvement and no major side effects. This suggests that weekly Isotretinoin could be a successful alternative for moderate acne in both males and females. To validate these findings, investigators propose a randomized controlled trial comparing weekly Isotretinoin to daily Doxycycline over four months. This study could confirm the safety and effectiveness of weekly Isotretinoin, as well as shed light on patient satisfaction, and long-term results compared to standard antibiotics. This research may offer a breakthrough in treating moderate acne while addressing concerns about antibiotic overuse.

DETAILED DESCRIPTION:
In current practice, treatment options for Moderate Acne Vulgaris remain limited. The mainstay of treatment remains long courses of oral antibiotics, mainly Tetracyclines. With the growing discussion of antibiotic stewardship, alternate and more effective therapies need to be explored. The efficacy of Isotretinoin, a Vitamin A derivative, for the treatment of Acne, has been well-established, but its use is often limited to treatment of severe Acne due to its possible side effects and standard lab monitoring. Several studies have explored low-dose Isotretinoin for Mild-to- Moderate Acne with promising results, however, to our knowledge, the first study looking at weekly dosing of Isotretinoin was conducted at our institution. In this proof-of-concept study, results showed improvement of Acne in almost all patients with no significant lab abnormalities or adverse events. Investigators concluded that weekly Isotretinoin dosing is a potential efficacious alternative for the treatment of Moderate Acne in both males and females and suggested study replication with a larger population and with comparison to standard of care (SOC) treatments. For these reasons, Investigators propose a randomized controlled trial comparing the efficacy of once weekly oral Isotretinoin dosing preceded by a 5-day daily loading dose to daily oral Doxycycline over a 4-month treatment period. This study has the potential to confirm the safety and efficacy of weekly dosed Isotretinoin for Moderate Acne treatment and highlight its adverse event profile, clinical effectiveness, patient satisfaction, and degree of sustained treatment response after drug cessation in comparison to standard of care Tetracyclines.

ELIGIBILITY:
Inclusion Criteria:

- Male and Female patients, 12 years and older with a diagnosis of Moderate Acne Vulgaris

Exclusion Criteria:

* Patients who are at baseline on long-term Tetracycline antibiotics, long-term Trimethoprim-Sulfamethoxazole, or on Spironolactone for any reason
* Patients who have taken Isotretinoin in the past 6 months
* Patients with hypersensitivity to Isotretinoin or to any of its components
* Females who are pregnant, likely to become pregnant, or will be breast-feeding during the study period
* Patients with a history of major depression, mania, or psychosis with an active episode during the past year including current psychotic symptoms and/or current suicidal ideation
* Adult patients with cognitive impairment
* Patients with baseline kidney or liver disease
* Patients with baseline hypertriglyceridemia
* Patients with history of or current pseudotumor cerebri
* Patients with any clinically significant unstable medical condition which could pose a risk to the safety of the patient
* Inability or unwillingness of subject or legal guardian/representative to give informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy using Comprehensive Acne Severity Scale | 10 months
  Determine the efficacy of weekly isotretinoin therapy for the treatment of moderate acne vulgaris compared to the current SOC therapy, systemic tetracyclines.

SECONDARY OUTCOMES:
Adverse Effect Questionnaire for isotretinoin | 4 months
  Compare the adverse effect profiles of weekly isotretinoin and SOC systemic tetracyclines when used for treatment of acne vulgaris. The questionnaire is written by study members asking patients if they experienced common side effects known to either medication.
Adverse Effect Questionnaire for SOC tetracycline | 4 months
  Compare the adverse effect profiles of weekly isotretinoin and SOC systemic tetracyclines when used for treatment of acne vulgaris. The questionnaire is written by study members asking patients if they experienced common side effects known to either medication.
Adverse Effects using Lipid Panel | 4 months
  Compare the adverse effect profiles of weekly isotretinoin and SOC systemic tetracyclines when used for treatment of acne vulgaris. Specifically the incidence of elevated triglycerides and elevated cholesterol will be recorded both based on the physiologic parameters measured in mg/dL.
Adverse Effects using Liver Function Test | 4 months
  Compare the adverse effect profiles of weekly isotretinoin and SOC systemic tetracyclines when used for treatment of acne vulgaris. Specifically the incidence of elevated alanine transaminase and elevated aspartate transaminase will be recorded both based on the physiologic parameters measured in IU/L.
Adverse Effects using Creatine phosphokinase | 4 months
  Compare the adverse effect profiles of weekly isotretinoin and SOC systemic tetracyclines when used for treatment of acne vulgaris. Specifically the incidence of elevated creatine phosphokinase will be recorded based on the physiologic parameters measured in IU/L.
Patient satisfaction using Dermatology Life Quality Index scale | 10 months
  Discern patient satisfaction with weekly isotretinoin or SOC systemic tetracyclines for acne treatment. Minimum score is 0, maximum score is 30. The higher the score the more patient quality of life is impaired.
Maintenance of treatment efficacy using Comprehensive Acne Severity Scale | 10 months
  Determine length of sustained treatment response after cessation of weekly isotretinoin or SOC systemic tetracycline therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Richmond, MD, MSCR, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States